CLINICAL TRIAL: NCT03124277
Title: A Whey Protein-based Nutritional Supplement Enriched in Vitamin D, Leucine and Calcium for Patients With Parkinsonism Undergoing Rehabilitation Treatment: a Randomized Trial
Brief Title: Nutritional Support for Rehabilitation In Parkinsonism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emanuele Cereda (Other)
Collaborators: ASST Gaetano Pini-CTO (Other); U.S. Riabilitazione Parkinson, Fondazione Gaetano e Piera Borghi di Brebbia (Unknown); Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor-Investigator, Emanuele Cereda, Co-Project Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 184_2017
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Disability Physical
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fortifit® (Experimental): Best local diet + two servings (40 grams each) of powder (Fortifit®; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Interventions: Dietary Supplement: Fortifit®
- Control group (Other): Best local diet
  Interventions: Other: Control Group

INTERVENTIONS:
Dietary Supplement: Fortifit® — Best local diet + two servings (40 grams each) of powder (Fortifit®; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Arms: Fortifit®
Other: Control Group — Best local diet
  Arms: Control group

SUMMARY:
This randomized, trial will tested the hypothesis that nutritional supplementation with whey protein, essential amino acids - mainly leucine - vitamin D and calcium would increase the efficacy of physical rehabilitation in old adults suffering from Parkinson's disease o parkinsonism

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease o parkinsonism
* admission for physical rehabilitation
* Informed consent

Exclusion Criteria:

* Any malignant disease during the last five years
* Known kidney failure (previous glomerular filtration rate <30 ml/min);
* Known liver failure (Child B or C)
* Psychiatric disease
* Endocrine disorders associated with disorders of calcium metabolism (excluding osteoporosis)
* Indications related to the study product:

More than 10 μg (400 IU) of daily Vitamin D intake from medical sources More than 500 mg of daily calcium intake from medical sources. Adherence to a high energy or high protein diet up or use of protein containing or amino acid containing nutritional supplements up to three months before starting the study.

* Known allergy to milk, milk products or other components of the proposed interventions
* Indication to or ongoing artificial nutrition support
* Inclusion in other nutrition intervention trials
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Functional status - distance walked during the six minutes walking test | 30 days
  Change in the distance walked during the six minutes walking test

SECONDARY OUTCOMES:
Functional status - timed up and go test | 30 days
  Change in timed up and go test
Functional status - Berg balance scale | 30 days
  Change in Berg balance scale score
Functional status - handgrip strength | 30 days
  Change in handgrip strength
Functional status - gait speed | 30 days
  Change in gait speed (4 minutes walking test)
Self-perceived functional status | 30 days
  Change in Self-assessment Parkinson's Disease Disability Scale
Body weight | 30 days
  Change in body weight
Muscle mass | 30 days
  Change in muscle mass
Adverse events | 30 days
  Occurrence of adverse events
Treatment continuation | 30 days
  Likelihood that patients would continue taking the trial treatment as assessed by a self-rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Michela Barichella, MD, Principal Investigator — Centro Parkinson, ASST Gaetano Pini-CTO di Milano
Locations (1):
- Centro Parkinson, ASST Gaetano Pini-CTO, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barichella M, Cereda E, Pinelli G, Iorio L, Caroli D, Masiero I, Ferri V, Cassani E, Bolliri C, Caronni S, Maggio M, Ortelli P, Ferrazzoli D, Maras A, Riboldazzi G, Frazzitta G, Pezzoli G. Muscle-targeted nutritional support for rehabilitation in patients with parkinsonian syndrome. Neurology. 2019 Jul 30;93(5):e485-e496. doi: 10.1212/WNL.0000000000007858. Epub 2019 Jul 5. PMID 31278117